CLINICAL TRIAL: NCT03972202
Title: The Role of Cerebellum in Speech
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Berkeley (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 19-27146; 1R01DC017091-01A1 (NIH)
Record Dates: First submitted 2019-05-24; First posted 2019-06-03 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Cerebellar Ataxia; Dysarthria; Healthy
Keywords: dysarthria; ataxia; cerebellum; cerebellar; adult; speaking; language; TMS; MRI; speech
MeSH Terms: conditions — Cerebellar Ataxia; Dysarthria; Ataxia; Speech; Language | interventions — Magnetic Resonance Imaging; Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Patients with cerebellar ataxia (CA) (Experimental): Behavioral testing including various speaking tasks Magnetic resonance imaging (MRI)
  Interventions: Diagnostic Test: MRI; Behavioral: Speech-motor behavioral testing
- Matched controls (Active Comparator): Behavioral testing including various speaking tasks Magnetic resonance imaging (MRI)
  Interventions: Diagnostic Test: MRI; Behavioral: Speech-motor behavioral testing
- Additional healthy volunteers (Experimental): Behavioral testing including various speaking tasks Magnetic resonance imaging (MRI) Transcranial magnetic stimulation (TMS)
  Interventions: Diagnostic Test: MRI; Device: TMS; Behavioral: Speech-motor behavioral testing

INTERVENTIONS:
Diagnostic Test: MRI — Brain MRI will be performed (no contrast) to correlate brain anatomy/function with behavioral testing.
  Other Names: Magnetic Resonance Imaging
Device: TMS — Repetitive TMS will be applied to transiently disrupt cerebellar speech pathways.
  Other Names: Transcranial Magnetic Stimulation; Repetitive TMS; rTMS
  Arms: Additional healthy volunteers
Behavioral: Speech-motor behavioral testing — Language/speaking tasks will be performed during which participants are asked to speak in response to audio/video cues; participants' responses will be recorded. For patients with cerebellar ataxia, additional diagnostic surveys may be completed.

SUMMARY:
This study will investigate the how the cerebellum is involved in speech motor learning over time and short-term corrections in patients with cerebellar ataxia and healthy controls. This will be accomplished through three approaches: behavioral studies, magnetic resonance imaging (MRI), and transcranial magnetic stimulation (TMS). During behavioral studies, participants will be asked to speak into a microphone while their voice is played back over earphones, and to do other speaking tasks. MRI will be acquired to perform a detailed analysis on brain function and anatomy related to speech and the cerebellum. In healthy controls, TMS will also be performed to temporarily disrupt the cerebellum before, during, or after the participant performs speaking tasks. Patients with cerebellar ataxia and healthy volunteers will be asked to complete behavioral studies and/or MRI; healthy volunteers may be asked to additionally participate in TMS.

DETAILED DESCRIPTION:
This study will investigate the role of the cerebellum in speech, building upon prior work in understanding cerebellar function in reaching and walking. Neuroimaging and lesion studies have provided strong evidence that the cerebellum is an integral part of the speech production network, though its precise role in the control of speech remains unclear. Furthermore, damage to the cerebellum (either degenerative or focal) can lead to ataxic dysarthria, a motor speech disorder characterized, in part, by impaired articulation and severe temporal deficits. This project seeks to bridge the gap between theoretical models of cerebellar function and the speech symptoms associated with ataxic dysarthria. Two mechanisms underlie speech motor control - feedback and feedforward control. In feedback control, speakers use sensory feedback (e.g., of their own voice) to control their speech. In feedforward control, speakers use knowledge gained from their past speech productions, rather than on-line feedback, to control their speech. This study entails a systematic plan to elucidate the role of the cerebellum in feedforward and feedback control of speech. A central hypothesis is that the cerebellum is especially critical in the feedforward control of speech, but has little involvement in feedback control. To explore this hypothesis, we will obtain converging evidence from three innovative methodologies: 1) Neuropsychological studies of speech-motor responses to real-time altered auditory feedback in patients with cerebellar atrophy (CA) and matched healthy controls, 2) Parallel studies in healthy controls undergoing theta-burst transcranial magnetic stimulation to create "virtual lesions" of the cerebellum, and 3) Structural and functional studies in CA patients to examine the relationship between cerebellar lesion location, dysarthria symptoms, and feedforward and feedback control ability.

Speech provides an important opportunity to examine how well current theories of cerebellar function generalize to a novel effector (vocal tract) and sensory (auditory) domain. Its purpose for communication imposes exacting spectro-temporal constraints not seen in other motor domains. Furthermore, the distinctive balance of feedback and feedforward control in speech allows us to examine changes in both control types subsequent to cerebellar damage. Critically, this is the first work examining the link between theoretically motivated control deficits in CA patients and the speech symptoms associated with ataxic dysarthria, as well as their neural correlates.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of cerebellar ataxia (CA) resulting from degeneration of the cerebellum AND normal hearing abilities OR
* Healthy volunteers with no known history of physical or neurological abnormalities AND normal speech, hearing, and reading abilities
* For some studies, primary language of American English may be required

Exclusion criteria for healthy volunteers:

* Neurological impairment or psychiatric illness

Exclusion criteria for participants with cerebellar ataxia (CA):

* Neurological impairment or psychiatric illness apart from those arising from cerebellar damage

Exclusion criteria for participants with CA or for healthy volunteers participating in MRI (may still be eligible for other study procedures):

* Any contraindication to participating in an MRI study including the following: implanted metallic parts or implanted electronic devices, including pacemakers, defibrillators, stimulators, or implant medication pump, or nonremovable piercings; aneurysm clip or other metal in the head (except mouth); claustrophobia precluding MRI

Exclusion criteria for healthy volunteers participating in TMS (may still be eligible for other study procedures):

* Any contraindications to participating in a TMS study including the following: epilepsy, use of certain medications, heart disease, and pregnancy; scalp wounds or infections; any other contraindication discovered during screening procedures
* Any contraindication to participating in an MRI study including the following: implanted metallic parts or implanted electronic devices, including pacemakers, defibrillators, or implant medication pump, or nonremovable piercings; claustrophobia precluding MRI

Exclusion criteria for all potential participants:

* Pregnant or trying to become pregnant (may still be eligible for behavioral studies only)
* History of alcohol abuse, illicit drug use or drug abuse or significant mental illness
* Hypertensive or hypotensive condition
* Any condition that would prevent the subject from giving voluntary informed consent
* Enrolled or plans to enroll in an interventional trial during this study
* Ongoing seizures that are not well controlled despite medication
* Use of hearing aid or other device to improve hearing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Speech-motor response percent compensation | Baseline
  Percent compensation is calculated as the following ratio: -100*(change in acoustic feature produced by the subject)/(change in acoustic feature caused by auditory feedback alteration). The negative sign ensures that changes produced by the subject that oppose the auditory feedback alteration changes are counted as positive compensation. Acoustic features used to compute percent compensation depend on the experiment performed and will include pitch or formant frequencies of subjects' output speech (measured by frequency in Hz), voice onset time (measured in milliseconds), fricative consonant duration (measured in milliseconds), and formant transition time (measured in milliseconds). We will look for short-term (within-trial) and long-term (across-trial) changes in percent compensation produced by subjects in response to alterations in subjects' auditory feedback they hear while speaking.
Dysarthria symptoms | Baseline
  Ataxic dysarthria (AD) symptoms will be quantified in patients with cerebellar ataxia (CA) by licensed speech-language pathologists using the Bogenhausen Dysarthria Scales (BoDyS), a dysarthria assessment tool that has been shown to be objective, reliable, and sensitive to dysarthria subtypes 31, 60, and 61. The BoDyS test entails 33 separate component ratings, including symptoms that may be related to feedforward and feedback components of speech motor control systems.
Voxel-based morphometry (VBM) | Baseline
  VBM will be applied to explore the functional organization of the cerebellum for speech production, focusing on psychophysical measures of speech motor control as well as clinical measures of dysarthric speech symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: John F. Houde, Ph.D., Principal Investigator — University of California, San Francisco; Srikantan S. Nagarajan, Ph.D., Principal Investigator — University of California, San Francisco; Richard Ivry, Ph.D., Principal Investigator — University of California, Berkeley; Ben Parrell, Ph.D., Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - University of California, Berkeley, Berkeley, California
  - University of California, San Francisco, San Francisco, California
  - University of Wisconsin--Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang EF, Niziolek CA, Knight RT, Nagarajan SS, Houde JF. Human cortical sensorimotor network underlying feedback control of vocal pitch. Proc Natl Acad Sci U S A. 2013 Feb 12;110(7):2653-8. doi: 10.1073/pnas.1216827110. Epub 2013 Jan 23. PMID 23345447
- [Background] Hinkley LB, Marco EJ, Brown EG, Bukshpun P, Gold J, Hill S, Findlay AM, Jeremy RJ, Wakahiro ML, Barkovich AJ, Mukherjee P, Sherr EH, Nagarajan SS. The Contribution of the Corpus Callosum to Language Lateralization. J Neurosci. 2016 Apr 20;36(16):4522-33. doi: 10.1523/JNEUROSCI.3850-14.2016. PMID 27098695
- [Background] Kort NS, Cuesta P, Houde JF, Nagarajan SS. Bihemispheric network dynamics coordinating vocal feedback control. Hum Brain Mapp. 2016 Apr;37(4):1474-85. doi: 10.1002/hbm.23114. Epub 2016 Feb 25. PMID 26917046
- [Background] Ranasinghe KG, Gill JS, Kothare H, Beagle AJ, Mizuiri D, Honma SM, Gorno-Tempini ML, Miller BL, Vossel KA, Nagarajan SS, Houde JF. Abnormal vocal behavior predicts executive and memory deficits in Alzheimer's disease. Neurobiol Aging. 2017 Apr;52:71-80. doi: 10.1016/j.neurobiolaging.2016.12.020. Epub 2017 Jan 3. PMID 28131013
- [Background] Moberget T, Gullesen EH, Andersson S, Ivry RB, Endestad T. Generalized role for the cerebellum in encoding internal models: evidence from semantic processing. J Neurosci. 2014 Feb 19;34(8):2871-8. doi: 10.1523/JNEUROSCI.2264-13.2014. PMID 24553928
- [Background] Sokolov AA, Miall RC, Ivry RB. The Cerebellum: Adaptive Prediction for Movement and Cognition. Trends Cogn Sci. 2017 May;21(5):313-332. doi: 10.1016/j.tics.2017.02.005. Epub 2017 Apr 3. PMID 28385461
- [Background] Koch G, Oliveri M, Torriero S, Salerno S, Lo Gerfo E, Caltagirone C. Repetitive TMS of cerebellum interferes with millisecond time processing. Exp Brain Res. 2007 May;179(2):291-9. doi: 10.1007/s00221-006-0791-1. Epub 2006 Dec 5. PMID 17146647
- [Background] Jenkinson N, Miall RC. Disruption of saccadic adaptation with repetitive transcranial magnetic stimulation of the posterior cerebellum in humans. Cerebellum. 2010 Dec;9(4):548-55. doi: 10.1007/s12311-010-0193-6. PMID 20665254
- [Background] Parrell B, Agnew Z, Nagarajan S, Houde J, Ivry RB. Impaired Feedforward Control and Enhanced Feedback Control of Speech in Patients with Cerebellar Degeneration. J Neurosci. 2017 Sep 20;37(38):9249-9258. doi: 10.1523/JNEUROSCI.3363-16.2017. Epub 2017 Aug 23. PMID 28842410
- [Background] Parrell, B., Agnew, Z., Houde, J., Nagarajan, S., & Ivry, R. (2016) Individuals with cerebellar degeneration correct for within-category variation of vowels even in the absence of auditory feedback. Talk presented at Society for Neuroscience 2016, San Diego, CA, November 2016.
- [Background] Parrell, B. (2017). Evidence for reward learning in speech production. Poster presented at the 7th International Conference on Speech Motor Control, Groningen, the Netherlands, July 2017.
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Oberman L, Edwards D, Eldaief M, Pascual-Leone A. Safety of theta burst transcranial magnetic stimulation: a systematic review of the literature. J Clin Neurophysiol. 2011 Feb;28(1):67-74. doi: 10.1097/WNP.0b013e318205135f. PMID 21221011
- [Background] Tarapore PE, Picht T, Bulubas L, Shin Y, Kulchytska N, Meyer B, Berger MS, Nagarajan SS, Krieg SM. Safety and tolerability of navigated TMS for preoperative mapping in neurosurgical patients. Clin Neurophysiol. 2016 Mar;127(3):1895-900. doi: 10.1016/j.clinph.2015.11.042. Epub 2015 Dec 11. PMID 26762952
- [Background] Tarapore PE, Picht T, Bulubas L, Shin Y, Kulchytska N, Meyer B, Nagarajan SS, Krieg SM. Safety and tolerability of navigated TMS in healthy volunteers. Clin Neurophysiol. 2016 Mar;127(3):1916-8. doi: 10.1016/j.clinph.2015.11.043. Epub 2015 Dec 11. No abstract available. PMID 26762949
- [Background] Wassermann EM. Side effects of repetitive transcranial magnetic stimulation. Depress Anxiety. 2000;12(3):124-9. doi: 10.1002/1520-6394(2000)12:33.0.CO;2-E. PMID 11126186
- [Background] Tarapore PE, Findlay AM, Honma SM, Mizuiri D, Houde JF, Berger MS, Nagarajan SS. Language mapping with navigated repetitive TMS: proof of technique and validation. Neuroimage. 2013 Nov 15;82:260-72. doi: 10.1016/j.neuroimage.2013.05.018. Epub 2013 May 20. PMID 23702420
- [Background] Tarapore PE, Tate MC, Findlay AM, Honma SM, Mizuiri D, Berger MS, Nagarajan SS. Preoperative multimodal motor mapping: a comparison of magnetoencephalography imaging, navigated transcranial magnetic stimulation, and direct cortical stimulation. J Neurosurg. 2012 Aug;117(2):354-62. doi: 10.3171/2012.5.JNS112124. Epub 2012 Jun 15. PMID 22702484